CLINICAL TRIAL: NCT06177548
Title: Safety and Efficacy of the Minimally Invasive Bentall Procedure Via a Small Right Intercostal Incision in Patients With Aortic Root Lesions: an Investigator-initiated, Single-center, Retrospective Cohort Study
Brief Title: Safety and Efficacy of the Minimally Invasive Bentall Procedure Via a Small Right Intercostal Incision in Patients With Aortic Root Lesions
Acronym: Mini-Bentall
Status: Recruiting | Type: Observational
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF2023LSK-434
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-03

CONDITIONS: Aortic Dissection; Aortic Root Aneurysm; Minimally Invasive Surgical Procedures
MeSH Terms: conditions — Aortic Dissection; Aortic Root Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Minimally invasive Group: Patients who underwent minimally invasive Bentall procedure will be included. The minimally invasive Bentall procedure is performed through a small incision in the right intercostal space.
  Interventions: Procedure: Minimally invasive Bentall procedure
- Control Group: Patient who underwent Bentall procedure through median sternotomy will be included.

INTERVENTIONS:
Procedure: Minimally invasive Bentall procedure — The minimally invasive Bentall procedure is performed through a small incision in the right intercostal space.
  Groups: Minimally invasive Group

SUMMARY:
This study intends to include patients who had aortic root lesions and were treated with Bentall surgery from January 2019 to July 2023 in the First Affiliated Hospital of Xi'an Jiaotong University. The patients will be divided into the minimally invasive group and control group according to the surgical methods: the former underwent minimally invasive Bentall surgery through a small right intercostal incision; the latter underwent traditional Bentall surgery through a median sternal incision. By comparing the clinical data of patients in two groups, we will investigate the effect and safety of minimally invasive Bentall surgery.

ELIGIBILITY:
Inclusion Criteria:

- Patients who were diagnosed with aortic root lesions and treated with the Bentall procedure at the First Affiliated Hospital of Xi'an Jiaotong University from January 2019 to July 2023 will be included in this study.

Exclusion Criteria:

* Previous sternotomy or aortic root surgery;
* Combined coronary artery disease requiring simultaneous coronary revascularization;
* Combined aortic arch lesions requiring simultaneous aortic arch surgery;
* Preoperative comorbidities with severe single or multiple organ failure;
* Incomplete clinical information;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were diagnosed with aortic root lesions and treated with the Bentall procedure at the First Affiliated Hospital of Xi'an Jiaotong University from January 2019 to July 2023 will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2023-12-11 (Actual); Primary Completion 2024-10-25 (Estimated); Study Completion 2024-12-28 (Estimated)

PRIMARY OUTCOMES:
30-day mortality rate | 1-month after the operation.
  It focuses on the mortality rate of all patients after the operation after 30 days. The data will be obtained from medical records.

SECONDARY OUTCOMES:
Mortality rate during hospitalization | About 10 days after the operation.
  It focuses on the mortality rate of all patients after the operation during hospitalization. The data will be obtained from medical records.
Blood transfusion volume during hospitalization | About 10 days after the operation.
  It focuses on the blood transfusion volumes of all patients after the operation during hospitalization. The data will be obtained from medical records.
Postoperative ICU length of stay | About 3 days after the operation.
  It focuses on the ICU length of stay of all patients after the operation. The data will be obtained from medical records.
Postoperative ventilation time | About 1 day after the operation.
  It focuses on the postoperative ventilation time of all patients after the operation. The data will be obtained from medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Yang Yan, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi'an Jiantong University, Xi'an, Shaanxi, China